CLINICAL TRIAL: NCT03883659
Title: Smartphone-based Mobility Assessment and Individualized Exercise Programs for Patients With Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wen-Hsu Sung, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FStraining
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Frozen Shoulder
Keywords: frozen shoulder; smartphone; home exercise program; range of motion
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: one assessor who don't know the group will measure the range of motion by using goniometer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional paper hangouts group (Active Comparator): patients use the traditional paper hangouts to conduct the home exercise program at home
  Interventions: Other: traditional paper hangouts
- smartphone group (Experimental): patients use the smartphone to conduct the home exercise program at home
  Interventions: Other: Smartphone

INTERVENTIONS:
Other: Smartphone — patients with frozen shoulder in the smartphone group will use the smartphone to conduct the home exercise program. The patients will be asked to follow the description to have mobility assessment at least 1 week and do the individualized exercise themselves.
  Arms: smartphone group
Other: traditional paper hangouts — patients with frozen shoulder in the smartphone group will use the paper hangouts to conduct the home exercise program. The content of the paper hangouts were description of the home exercise.
  Arms: traditional paper hangouts group

SUMMARY:
This study was to investigate the reliability and validity of the smartphone goniometer app to measure shoulder ROM in a modified position for patients with frozen shoulder, and compare the intervention effect and adherence to home exercise between the smartphone and traditional paper hangouts.

DETAILED DESCRIPTION:
This study was to investigate the reliability and validity of the smartphone goniometer app to measure shoulder ROM in a modified position for patients with frozen shoulder, and compare the intervention effect and adherence to home exercise between the smartphone and traditional paper hangouts. The outcome measure including shoulder range of motion, pain condition, home exercise adherence and satisfaction of smartphone program

ELIGIBILITY:
Inclusion Criteria:

* gradual shoulder pain and stiffness at least 4 months
* loss of active and passive shoulder mobility, shoulder external rotation <45 degree
* ability to use the smartphone

Exclusion Criteria:

* normal shoulder mobility
* diagnostic shoulder osteoarthritis
* nerve pain
* injection of corticosteroids in 3 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
home exercise adherence | 4 weeks
  the days patients do the home exercise program

SECONDARY OUTCOMES:
shoulder range of motion | baseline, 4 weeks
  the mobility of shoulder
Visual analog scale (VAS) | baseline, 4 weeks
  Ranged form 0 (minimum score) to 10 (Maximum score) ,the higher score represent more painful
System usability scale (SUS) | 4 weeks
  the satisfaction scale of the smartphone program

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hsu Sung, PhD, Principal Investigator — Principal Investigator
Locations (2):
- Taiwan (2):
  - Tri-Service General Hospital, Taipei, Neihu District
  - Yang Ming university, Taipei

IPD SHARING:
Plan to Share IPD: No